CLINICAL TRIAL: NCT03313388
Title: The Effect of Tart Cherry Juice on Fat Metabolism, Exercise Performance, and Recovery
Brief Title: Tart Cherry Juice for Exercise Performance and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 16-273
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Muscle Damage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tart Cherry Juice (Experimental): 290 mL per day of Tart Cherry juice for 7 days
  Interventions: Dietary Supplement: Drink
- Gatorade (Active Comparator): 290 mL per day of Gatorade for 7 days
  Interventions: Dietary Supplement: Drink

INTERVENTIONS:
Dietary Supplement: Drink — Beverage to be consumed

SUMMARY:
This study evaluates the effects of tart cherry juice consumption on endurance exercise performance, fat metabolism during exercise, blood pressure, and recovery from exercise as assessed by muscle pain, muscle strength and electrical properties of muscle. Comparisons will be made to Gatorade consumption. Participants include those who are moderately active and have experience with cycling.

DETAILED DESCRIPTION:
Tart cherries are rich in bioactive components (i.e. flavonoids) that have anti-inflammatory and anti-oxidant properties. Inflammation and lipid peroxidation causes damage of skeletal muscle membranes during intense exercise. The damage of muscle increases the amount of time for muscle to recover from intense exercise, and can cause muscle strength to be reduced for days. When tart cherries in a concentrated form (i.e. as juice or powder) are consumed in the days leading up to intense exercise, there is a protective effect against inflammation, and lipid peroxidation . This theoretically prevents damage to the lipid component of muscle fibre membranes and helps to preserve muscle function - when muscle is damaged by intense exercise (i.e. either repetitive aerobic activity or high-force muscle contraction), consumption of cherry juice enhances the rate of muscle strength recovery following exercise compared to when a placebo (i.e. non-cherry) beverage is consumed . Muscle damage may be protected by cherry juice consumption; however, all studies evaluating the protective effect of cherries have assessed muscle damage by measuring muscle proteins in the blood. This rather indirect measure of muscle damage is highly variable and not always an accurate assessment of muscle damage; this may be why some studies indicate a reduction in markers of muscle damage with cherry juice consumption while others do not.

A more direct assessment of muscle damage can be obtained by applying electrical stimulation at different frequencies to a muscle before and after intense exercise and assessing the reduction in force output in response to low-frequency and high-frequency stimulation. After intense exercise, the force output at low frequencies of stimulation is often reduced, while the force output at high frequencies is maintained; a phenomenon termed "low frequency fatigue". When muscle is stimulated to contract (either voluntarily by the nervous system or involuntarily through electrical stimulation) calcium is released inside muscle. This calcium release leads to muscle contraction. When muscle undergoes intense exercise, there is damage to muscle membranes, including membranes inside muscle that are responsible for calcium release. This causes a lower amount of calcium to be released with each muscle contraction. Normally, if high frequencies of electrical stimulation are applied to muscle, a very large amount of calcium is released inside muscle - an amount which is "more than enough" to cause a high amount of muscle contraction and high force output. If muscle fibre membranes responsible for release of calcium are damaged, a lower amount of calcium is released, but because "more than enough" calcium is usually released with high frequency stimulation, the lower amount of calcium released with muscle damage is still enough to cause high force of muscle contraction. The force response to low frequencies of stimulation; however, is dramatically reduced when muscle is damaged - usually only a small amount of calcium is released when low frequencies of stimulation are delivered to muscle. Following muscle damage, the smaller amount of calcium released causes lower force production at low stimulation frequency. Low force production at low stimulation frequencies, with a relatively maintained force production at high stimulation frequencies therefore indicates that muscle damage has occurred. This lower muscle force capability at low frequencies of stimulation has dramatic effects on endurance performance because typical endurance performance relies on repeated low-force muscle contractions, as opposed to the few high-force contractions that might be required in other sports (i.e. short sprinting events or field events such as shot put).

The study we are proposing will use this measurement (i.e. ratio of low frequency force to high frequency force output) as a more direct measure of muscle damage. We predict that if cherry juice is consumed in the days leading up to a bout of muscle-damaging endurance exercise, muscle damage will be lower (as indicated by a faster recovery of low-frequency fatigue following the bout of exercise) than when a comparison-drink (i.e. Gatorade) is consumed.

ELIGIBILITY:
Inclusion Criteria:

* experienced cyclist (i.e. bicycle exercise at a vigorous intensity on a regular basis)

Exclusion Criteria:

* Allergies to cherries

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Time time performance | Day 5 of beverage consumption
  Time to complete 10 km of cycling

SECONDARY OUTCOMES:
Fat oxidation | Day 5 of beverage consumption
  Fat oxidation determined from gas analysis
Carbohydrate oxidation | Day 5 of beverage consumption
  Carbohydrate oxidation determined from gas analysis
Blood pressure | Day 5 of beverage consumption
  Blood pressure assessed by continuous blood pressure monitor
Muscle pain | Change from baseline to before, and immediately, 24 hours, and 48 hours after exercise
  Muscle pain determined by a visual analog scale (participant marks a scale from 0 to 100 mm. A score of 0 mm is "no pain". A score of 100 mm is maximal pain).
Quadriceps strength | Change from baseline to before, and immediately, 24 hours, and 48 hours after exercise
  Knee extensor strength determined by isometric contraction
Low frequency fatigue | Change from baseline to before, immediately, 24 hours, and 48 hours after exercise
  Measured by force production at low and high stimulation frequencies as an index of muscle damage

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No